CLINICAL TRIAL: NCT01242150
Title: Noninvasive Continuous Positive Airway Pressure by Helmet or Facial Mask in Children: a Multicenter Randomized Controlled Study
Brief Title: Noninvasive Continuous Positive Airway Pressure (NCPAP) in Children
Acronym: NCPAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Prof. Pier Mannuccio Mannucci, Professor, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCHNN16011968
Record Dates: First submitted 2010-11-14; First posted 2010-11-16 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Acute Respiratory Failure
Keywords: Acute Respiratory Failure; Continuous Positive Airway Pressure; Infants; Helmet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NCPAP Helmet (Experimental): Infants with mild Acute Respiratory Failure who need NCPAP
  Interventions: Device: NCPAP by helmet
- NCPAP facial mask (Active Comparator): Infants with mild Acute Respiratory failure who need NCPAP
  Interventions: Device: NCPAP by facial mask

INTERVENTIONS:
Device: NCPAP by helmet — The infant helmet (Castar Starmed© Mirandola, Italy) is secured to a soft collar that adheres to the child's neck and is connected to a high flow NCPAP circuit (high fresh gas flow >40 L/min to avoid carbon dioxide rebreathing). To facilitate tolerance up to a maximum of 2 boluses of midazolam 0.1 mg/kg i.v. can be administered eventually followed by an i.v. continuous infusion rate according to OPS scale. Once the interface is positioned, a baseline Continuous Positive Airway Pressure (CPAP) level is set at 4 cm H2O and then raised in increments of 2 cm H2O every 20 min up to a maximum of 10 cm H2O. FiO2 is set to achieve a SpO2 ≥ 92%. If intolerance persisted despite sedative administration, the alternate interface can be used before considering tracheal intubation. All patients are kept in semirecumbent position.
  Other Names: Noninvasive Continuous Positive Airway Pressure by helmet
  Arms: NCPAP Helmet
Device: NCPAP by facial mask — The size of NCPAP full face or nasal masks are chosen to be more comfortable for the infants (Respironics, Murrysville). The masks are secured by head straps while avoiding a tight fit and air leaks. A protective hydrocolloid sheet was applied over the nasal bridge (DuoDERM, ConvaTec, Deeside, UK). After a short adaptation period, it is firmly applied on the face by a pediatric head cap (Respironics, Murrysville ) to minimize air leaks. The mask is then connected to the same circuit previously described for helmet NCPAP.
  Other Names: Noninvasive Continuous Positive Airway Pressure by mask
  Arms: NCPAP facial mask

SUMMARY:
In critically ill pediatric patients with Acute Respiratory Failure (ARF), Noninvasive Continuous Positive Airway Pressure (NCPAP) is applied to avoid intubation and all related complications such as tracheal injury and predisposition to nosocomial pulmonary infections. The choice of the interface is one of the crucial issues affecting treatment outcome in pediatric age and in particular in preschool children in whom intolerance frequently compromise noninvasive respiratory treatment. NCPAP is applied either through nasal or facial tight fitting masks and the most important principle in guiding the selection of an interface is that it should fit comfortably. However, while nasal mask can leak gas when the infant opens his/her mouth, facial mask can cause significant gastric distension and vomiting, with risk of aspirating gastric contents. Moreover, complications such as air leaks, skin irritation on the bridge of the nose, and discomfort reported with nasal or facial masks in children frequently lead to interruption of the respiratory treatment. Thus, improving the interface between the patient and the ventilator would be expected to facilitate longer and more effective application of NCPAP.

A new small helmet specifically designed for young infants has been recently introduced to administer NCPAP. In a recent short term crossover physiological randomized controlled trial, the investigators found that NCPAP by helmet was associated with enhanced feasibility, less need of sedation and prolonged application time (see references below). The purpose of this prospective randomized multicenter study is to compare the efficacy and feasibility of NCPAP delivered either by helmet or by facial mask to treat acute respiratory failure in infants admitted to Pediatric Intensive Care Unit (PICU).

DETAILED DESCRIPTION:
Prospective, randomized, multicenter clinical study on parallel groups involving all consecutive infants ageing >1 month <2 yrs, admitted to PICU at Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Children Hospital V. Buzzi Milan, and at Gemelli Università Cattolica del Sacro Cuore Rome, for mild to severe acute respiratory failure (ARF). For screening purposes ARF is defined as the presence of all the following: respiratory rate >50 breaths/min; Partial arterial Oxygen tension/Inspired Oxygen Fraction ratio (PaO2/FiO2) <300, chest x-ray compatible with clinical diagnosis, no significant clinical improvement after breathing oxygen at 8 l/min or more for at least 15 min.

Before enrollment patients receive standard medical therapy consisting of oxygen administration via Venturi mask to achieve a peripheral oxygen saturation (SpO2)> 92% and medications including aerosolized salbutamol or adrenaline, anticholinergic, steroids, intravenous antibiotics, correction of electrolytes, and intravascular volume abnormalities as clinically indicated. Heart rate, systemic arterial blood pressure, respiratory rate, and SpO2 are continuously monitored. Patients are defined as requiring NCPAP if they deteriorate despite medical treatment and meet at least one of the following criteria: SpO2<90% with FiO2 > 40%, arterial pH < 7.25, respiratory rate > 50 breaths/min, severe deterioration in mental status (Glasgow Coma Scale < 10). Eligible patients meeting two or more of the above criteria are randomly assigned to receive NCPAP either by full-face mask or by helmet. Random assignment is made by sealed envelopes. Informed consent is obtained from at least one parent or a legal guardian before the enrollment in the study.

To facilitate tolerance up to a maximum of 2 boluses of midazolam 0.1 mg/kg intravenous can be administered eventually followed by an intravenous continuous infusion rate, according to the attending physician's discretion. Once the interface is positioned, a baseline CPAP level is set at 4 cm H2O and then raised in increments of 2 cm H2O every 20 min up to a maximum of 10 cm H2O to improve respiratory performance as evidenced by oxygen need, respiratory rate decrease and the reduction of accessory muscles activity. Inspired Oxygen Fraction (FiO2) is set to achieve a SpO2≥ 92%. NCPAP is administered intermittently for at least 8 hours a day for the first 48 hours after enrollment, but the daily administration can last longer if well tolerated or less if either weaning or intubation criteria are achieved. In case of persistent intolerance to the interface despite sedative administration, the alternate interface can be used before considering tracheal intubation. For patients with a nasogastric tube a seal connector in the lower rigid part of the helmet or in the dome of the mask are used to avoid air leaks. All patients are kept in semirecumbent position.

Criteria for weaning NCPAP can be discontinued if infants show normal mental status, stable haemodynamics, SpO2>94% in room air and no activation of accessory muscles or paradoxical abdominal motion.

Criteria for endotracheal intubation The predetermined criteria for endotracheal intubation NCPAP administration, despite the use of NCPAP, any hemodynamic or electrocardiographic instability; inability to improve dyspnea, conditions requiring intubation either to protect the airways or to manage copious tracheal secretions.

End points and definitions The primary outcome variable is the rate of treatment failure in each group. Treatment failure is defined as infants either shifted to the alternate interface because of intolerance or tracheally intubated because of gas exchange deterioration. A successful treatment is defined as the ability to administer NCPAP for at least 8 hours a day for the first 24 hours and to avoid tracheal intubation in the first 48 hours. Secondary end-points included: gas exchange improvement, complications not present on admission, length of the stay and mortality in PICU.

Arterial partial oxygen and carbon dioxide tension, arterial pH, respiratory rate, heart rate and systolic arterial blood pressure are evaluated at 2, 24 and 48 hours after enrollment.

Early improvement in oxygenation is defined as an increase in PaO2/FiO2 > 20% above baseline; sustained improvement is defined as the ability to maintain increase in oxygenation at 24 hours after enrollment.

At the same time intervals Objective Pain Scale (OPS), an index of patient intolerance to the interface and Respiratory Effort Score (RES), an index of respiratory muscles activity, are recorded. Intolerance to the NCPAP treatments defined as an increment in OPS>4. In the first 24 hours the total amount of sedation and the total duration of NCPAP administration are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* PaO2/FiO2 ratio <300
* Respiratory rate >50 breaths/min
* Chest x-ray compatible with pulmonary infection
* No clinical improvement after breathing oxygen at 8 l/min or more for at least 15 min

Exclusion Criteria:

* Presence of an endotracheal tube or a tracheostomy before PICU admission
* Facial deformities
* Upper airway obstruction
* Cyanotic congenital heart disease
* Facial trauma
* Recurrent apnea
* Neuromuscular weakness
* Pulmonary hypoplasia
* Pulmonary vascular anomalies
* Imminent respiratory or cardiac arrest
* COPD and/or chronic CO2 retention
* Status asthmaticus
* Pneumothorax
* Hemodynamic instability
* Alteration in consciousness with a Glasgow coma score (GCS) <10
* Aspiration or excessive bronchial secretions
* Enrollment in other research protocol

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome variable is the number of treatment failure in each nCPAP group. | 1 year

SECONDARY OUTCOMES:
Gas exchange improvement | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Chidini, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (4):
- Italy (4):
  - Department of Anesthesia and Intensive Care, Vittore Buzzi Children's Hospital, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Department of Anesthesia and Intensive Care, Policlinico Gemelli, Rome
  - Department of the Environment, Healthy and Safety, University of Insubria, Varese

REFERENCES:
- [Result] Chidini G, Calderini E, Pelosi P. Treatment of acute hypoxemic respiratory failure with continuous positive airway pressure delivered by a new pediatric helmet in comparison with a standard full face mask: a prospective pilot study. Pediatr Crit Care Med. 2010 Jul;11(4):502-8. doi: 10.1097/PCC.0b013e3181b8063b. PMID 19794328
- [Result] Chidini G, Calderini E, Cesana BM, Gandini C, Prandi E, Pelosi P. Noninvasive continuous positive airway pressure in acute respiratory failure: helmet versus facial mask. Pediatrics. 2010 Aug;126(2):e330-6. doi: 10.1542/peds.2009-3357. Epub 2010 Jul 26. PMID 20660548